CLINICAL TRIAL: NCT00446823
Title: A Prospective, Randomized, Controlled Clinical Study to Evaluate the Effectiveness of a Cellulose Matrix Wound Dressing for Autolytic Debridement and Healing of Chronic Venous Ulcers
Brief Title: Effectiveness of XCell on Autolytic Debridement of Venous Ulcers
Acronym: XCell
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xylos Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XC-0201-VU
Record Dates: First submitted 2007-03-09; First posted 2007-03-13 (Estimated); Last update posted 2007-03-13 (Estimated); Status verified 2007-03

CONDITIONS: Venous Ulcer
Keywords: Wound healing; Venous stasis ulcer; Cellulose dressing; Gauze dressing; Chronic wound
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: XCell cellulose wound dressing
Device: Impregnated gauze dressing

SUMMARY:
This clinical trial is designed to evaluate the effect of XCell cellulose wound dressing for its ability to naturally (autolytically) remove nonviable tissue and create a healthy vascular wound bed. Results will compare venous ulcers treated with Xylos XCell cellulose dressing plus standard care to those treated with standard care alone. The hypothesis is that XCell will demonstrate more autolytic debridement than the standard of care.

DETAILED DESCRIPTION:
Chronic wounds are a problem for both the patient and the health care provider. The definition of a chronic wound is one that deviates from the expected sequence of repair in time, appearance and response to aggressive treatment. These wounds can be separated into distinct classes by etiology, specifically, pressure, ischemic, venous, neuropathic, diabetic, inflammatory or infective wounds. The degree of severity can be quite diverse spanning the range of superficial epidermal injury to full-thickness skin loss with extensive destruction, tissue necrosis, and damage to supporting structures including muscle, tendon, and or bone. Treatment of chronic wounds should begin with the management of the underlying etiology. For example: In pressure ulcers the elimination or reduction of pressure is the primary goal; In venous ulcers, improving venous insufficiency or reducing venous hypertension should come first; and in diabetic foot ulceration, proper off loading is essential. After treatment of the underlying pathology, one thing that all chronic wounds have in common is that they require wound bed preparation in order to stimulate the healing process.

Most clinical wound care trials to evaluate therapeutic agents for wounds have been designed to measure healing as the primary endpoint. The sequence of events begins with patient examination, wound classification and then the application of the test agent. In most cases, the test agent is placed over a wound that is contaminated with excessive bacteria, needs debridement, or requires wound bed preparation such as exudate control.

A new wound dressing (Xylos XCell cellulose wound dressing) is a unique biosynthetic matrix material that is hydrophilic and has excellent tensile strength. It has the ability to deliver moisture into a wound or absorb moisture. This cellulose matrix is microbially derived, biocompatible, pyrogen-free and completely non-toxic. In previous clinical trials this dressing displayed the ability to aid the natural process of autolytic wound debridement, cleansing and exudate control. From initial observations, it appears that this cellulose matrix provides an environment that prepares the wound bed by eliminating nonviable tissue, reducing bacterial burden, controlling exudate and exposing healthy granulation tissue. With successful wound bed preparation one can now concentrate on healing the chronic wound.

This clinical trial is designed to evaluate the natural cleansing (autolytic debridement process) and healing attributes of this new cellulose wound dressing compared to standard of care (impregnated gauze). Venous ulcers have been chosen as the model because these wounds are often covered with thick fibrous non-viable tissue, are poorly vascularized, are contaminated with numerous bacteria and exude copious amount of wound fluid.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any race and are between 18 and 90 years of age.
* Patients that are able to understand and are willing to give written informed consent.
* Patients that have a non-healing open venous ulcer for at least one month.
* Patients that have greater than 50% of the ulcers surface area covered with non-viable tissue such as fibrin slough, dry crust or a combination of both.
* Patients that have the clinical signs and symptoms of venous ulceration such as varicosities, hyper pigmentation, stasis dermatitis, lipodermatosclerosis, and edema.
* Patients that have a venous ulcer with a surface area of greater than or equal to 1.5 cm2.
* Patients that have an ankle to brachial index (ABI) > 0.70.

Exclusion Criteria:

* Study wound (target ulcer) etiology is other than venous insufficiency.
* Patient has peripheral arterial disease as determined by the following criteria: Ankle/Brachial Index < 0.7 (ulcerated leg), evidence of intermittent claudication.
* Patient has the presence of any of the following in the area of the ulcer: cellulitis, osteomyelitis, and ulcer with exposed bone, tendon or fascia.
* Patient has a known hypersensitivity to dressing components.
* Patient is receiving corticosteroids, immunosuppressive agents, radiation therapy, or chemotherapy where in the investigator's opinion could interfere with wound healing .
* Patient is known to have uncontrolled diabetes mellitus (as defined by the investigator).
* Patient is known to have immunodeficiency disorders that interfere with wound healing.
* Patient has a history of sickle cell anemia, thalassemia, vasculitis, rheumatoid arthritis, lupus erythematosus, polyarteritis nodosa, scleroderma or any connective tissue or collagen vascular disorder.
* Patient has wounds that have been treated with an investigational product within the past thirty days.
* Patient has not signed the informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2002-06; Study Completion 2003-12

PRIMARY OUTCOMES:
Ability of dressing to autolytically debride wound

SECONDARY OUTCOMES:
To evaluate and compare healing of wounds treated with XCell or control
To evaluate level of pain

CONTACTS AND LOCATIONS:
Overall Officials: Oscar M Alvarez, Ph.D., Principal Investigator — University Wound Clinics, LLC
Locations (3):
- United States (3):
  - Boston University School of Medicine, Boston, Massachusetts
  - University Wound Care Center, The Bronx, New York
  - Etris Associates, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Frankel VH, Serafica GC, Damien CJ. Development and testing of a novel biosynthesized XCell for treating chronic wounds. Surg Technol Int. 2004;12:27-33. PMID 15455308
- [Result] Alvarez OM, Patel M, Booker J, Markowitz L. Effectiveness of a biocellulose wound dressing for the treatment of chronic venous leg ulcers: Results of a single center randomized study involving 24 patients. WOUNDS 16(7):224-233, 2004